CLINICAL TRIAL: NCT06866730
Title: Effect of Intensive Repetitive Motor Training in Toy Manipulation Supported by Gamified Physical Training Software in Children and Adolescents with Neurological Disorders Impacting Motor Skills
Brief Title: Effect of Using an Object Handling Serious Game on Upper Limb Rehabilitation for Children with Neurological Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ellen Poidatz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REPLAY
Record Dates: First submitted 2024-11-18; First posted 2025-03-10 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Serious game upper limb rehabilitation (Experimental): 4 weeks program with 3 sessions per week of 40 minutes of serious game to improve upper limp motor function
  Interventions: Device: Serious game

INTERVENTIONS:
Device: Serious game — Serious game in which participants manipulate instrumented toys

SUMMARY:
Cerebral palsy, and more broadly neurological disorders, can lead to significant motor impairments that impact individuals' daily lives. To address these limitations, the French National Authority for Health has issued recommendations for rehabilitative care, highlighting intensive training programs, physical activity, and interactive computer games. Scientific literature has also demonstrated the benefits of therapies that incorporate repetition.

In this study, the investigators aimed to train patients in producing grasp-and-release movements, and more broadly *reach-to-grasp* actions, in a manner intensified by movement repetition. To mitigate the boredom inherent to such repetitive tasks, the invesigators developed a device resembling a serious game, equipped with software, a modular physical platform, and two instrumented figurines designed to interact with the software.

Intensive therapy through repetitive movements, supported by the engaging nature of serious games, is expected to improve the manual skills of children with neurological disorders causing motor impairments.

To test this hypothesis, a cohort of 5 to 10 children aged 4 to 17 years with neurological disorders causing motor impairments will be invited to participate in the protocol. Participants will first undergo a baseline assessment, which will include repeated measurements of their score on the *Box and Blocks Test* and the active range of motion (AROM) of the wrist in extension and supination. An *Assisting Hand Assessment (AHA)* test will also be conducted.

Following this, a 4-week intervention will be implemented, consisting of three 40-minute sessions per week. During these sessions, the child will play the game and complete the *Box and Blocks Test* as well as active range of motion assessments.

In total, approximately 4 hours of gameplay is estimated over the course of the intervention, which will conclude with a repeat of the AHA test.

A follow-up assessment will take place two months after the intervention's end, with a single measurement of the three parameters (*Box and Blocks Test*, AROM, and AHA).

ELIGIBILITY:
Inclusion Criteria:

* Neurological disorder causing motor impairment
* Age 4 to 17 years old
* MACS level I to III
* Ability to cooperate, understand, and follow simple instructions to play the game.
* Patient affiliated with the French social security system.
* Voluntary patient whose parents have given consent for their child to participate in the study.

Exclusion Criteria:

* A diagnosis of photosensitive epilepsy mentioned in the medical record AND/OR a note in the child's medical record or reported by the parents of a history of seizures triggered by video game use.
* Botulinum toxin treatment within the 3 months prior to the study or intensive rehabilitation of manual skills (e.g., mCIMT, HABIT, etc.).
* Sensory and/or cognitive impairments that would interfere with playing the game.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Box and Blocks test | 3 months
  Participant must transfer, one by one, with one hand, a maximum number of cubes from one side to the other of the box in 1 minute. A higher score represents better performance.

SECONDARY OUTCOMES:
Active Range of Motion | 3 months
  Measurement of the angle of active wrist extension and supination.
Assisting Hand Assessment | 3 months
  Determine a score of natural use of the affected upper limb in standardized activity test. The Assisting Hand Assessment contains 20 items rated on a 4-point scale (4=effective, 3=somewhat effective, 2=ineffective, and 1=does not do). A higher score therefore represents better performance.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CRMTP Elisatbeth de la Panouse-Debré, Antony
  - Fondation Ellen Poidatz, Saint-Fargeau-Ponthierry